CLINICAL TRIAL: NCT00250900
Title: Wait and See Antibiotic Prescription for Acute Otitis Media: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WASPYALE2005; #AI01703 NIH; #MO1-RR00125 GCRC
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2005-11

CONDITIONS: Otitis Media
Keywords: Otitis; Antibiotic; Prescription
MeSH Terms: conditions — Otitis Media; Otitis

INTERVENTIONS:
Behavioral: Prescription Fill Status

SUMMARY:
To determine if a wait and see prescription for ear infections in childhood reduces use of antibiotics compared to an immediate prescription

DETAILED DESCRIPTION:
We conducted a randomized, controlled trial evaluating a consecutive series of children diagnosed with AOM during a one year period in an urban pediatric emergency department, utilizing diagnostic recommendations from contemporary evidence-based guidelines. The objectives of the study were to determine whether treatment of AOM using a "Wait and See Prescription" (WASP) significantly reduces use of antimicrobials compared with a "Standard Prescription" (SP) and to evaluate the effects of this intervention on clinical symptoms and adverse outcomes related to antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 months - 12 years who were diagnosed with Acute Otitis Media

Exclusion Criteria:

* clinician suspicion or diagnosis of a concurrent bacterial infection
* patient appeared "toxic" as determined by the PEM clinician
* patient was hospitalized
* history of compromised immunity
* patient was treated with antimicrobials in the preceding seven days
* either tympanic membrane was perforated
* myringotomy tubes were present
* uncertain access to medical care
* primary language of the parent or guardian was neither English nor Spanish
* prior enrollment in the study

Ages: 6 Months to 12 Years | Sex: All
Age Groups: Child
Enrollment: 240
Dates: Start 2004-07; Study Completion 2005-08

PRIMARY OUTCOMES:
Proportion of each group that filled the antibiotic prescription

SECONDARY OUTCOMES:
Clinical course of the illness; side effects of medications; days of school/work missed; unscheduled medical visits

CONTACTS AND LOCATIONS:
Overall Officials: David M Spiro, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Result] Spiro DM, Tay KY, Arnold DH, Dziura JD, Baker MD, Shapiro ED. Wait-and-see prescription for the treatment of acute otitis media: a randomized controlled trial. JAMA. 2006 Sep 13;296(10):1235-41. doi: 10.1001/jama.296.10.1235. PMID 16968847